CLINICAL TRIAL: NCT04385849
Title: Phase 1b, Randomized, Blinded, Placebo-controlled Study of the Safety of Therapeutic Treatment With an Immunomodulary Agent (N-803 in Adults With COVID-19
Brief Title: Study of the Safety of Therapeutic Treatment With an Immunomodulatory Agent (N-803) in Adults With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QUILT-COVID-19
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ALT-803; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): N-803 Recombinant human super agonist interleukin-15 (IL-15) complex
  Interventions: Biological: N-803
- Placebo Arm (Placebo Comparator): Sterile saline solution
  Interventions: Other: Saline

INTERVENTIONS:
Biological: N-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: Experimental Arm
Other: Saline — Sterile saline solution
  Arms: Placebo Arm

SUMMARY:
This is a phase 1b, randomized, blinded, placebo-controlled study in adult subjects with COVID-19. This clinical trial is designed to assess the safety and immunostimulatory activity of N-803.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Has laboratory-confirmed positive novel coronavirus (SARS-CoV-2) test, as determined by polymerase chain reaction (PCR), or other commercial or public health assay in any specimen < 72 hours prior to enrollment, or meets the criteria to guide the evaluation and testing of patients under investigation (PUI) for COVID-19 (https://emergency.cdc.gov/han/2020/HAN00428.asp).
4. Has a confirmed NEW score of 0-5.
5. Has at least one of the following high-risk factors associated with a higher risk of COVID-19 progression:

   1. Age ≥ 60 years.
   2. Hypertension currently managed by at least 1 antihypertensive medication.
   3. Type 1 or 2 diabetes.
   4. Chronic obstructive pulmonary disease (COPD) diagnosed per medical history.
6. Adequate respiratory and heart function, evidenced by the following laboratory results:

   1. Respiratory rate (RR) < 20 breaths per minute (bpm).
   2. Heart rate (HR) < 90 beats per minute (bpm).
   3. Arterial oxygen saturation (SaO2) > 93% on room air.
7. Agrees to the collection of nasopharyngeal (NP) swabs and venous blood per protocol.
8. Ability to participate in required study visits and participate in adequate follow-up, as required by this protocol.
9. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception while on study and for at least 1 month after the last dose of N-803. Non-sterile male subjects must agree to use a condom while on study and for up to 1 month after the last dose of N-803. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), oral contraceptives, and abstinence.

Exclusion Criteria:

1. Shortness of breath or hypoxia defined by a ratio of partial pressure of arterial oxygen to the percentage of inspired oxygen (PaO2/FiO2) ≤ 300 mmHg or signs of serious lower airway disease.
2. Signs or symptoms of acute respiratory distress syndrome (ARDS), systemic inflammatory response syndrome (SIRS)/shock, or cardiac failure; or need for supplemental oxygen.
3. Inflammatory markers (C-reactive protein [CRP], lactate dehydrogenase [LDH], d-dimer, ferritin, and IL-6) > 1.5 × upper limit of normal (ULN).
4. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
5. Pregnant and nursing women. A negative serum or urine pregnancy test during screening prior to the first dose must be documented before N-803 is administered to a female subject of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Francis, Lynwood, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm | Placebo Arm
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the Placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Placebo Arm | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (0) |  | 70 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: AEs will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Time Frame: 3 days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm | Placebo Arm
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: The planned follow up time was 29 days post dose, but the one participant enrolled was lost to follow up 3 days post dose.
Description: The subject was on study for 3 days and lost to follow up. No adverse events were reported within those 3 days. No other subjects were enrolled.
Arm/Group | Experimental Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
The study is terminated early due to low enrollment. Effect of the study drug on efficacy was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT04385849/Prot_SAP_000.pdf